CLINICAL TRIAL: NCT04885543
Title: Observational Study of the Clinico-biological Evolution and the Standard of Care Offered to Symptomatic Covid-19 Patients in Sub-Saharan Africa
Brief Title: COVID-19 STAndard of Care in Sub-Saharan Africa
Acronym: COVISTA
Status: Completed | Type: Observational
Sponsor: Alliance for International Medical Action (Other)
Responsible Party: Sponsor
Other Study IDs: ALIMA02
Record Dates: First submitted 2021-05-06; First posted 2021-05-13 (Actual); Last update posted 2021-05-13 (Actual); Status verified 2021-05

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study was conducted in three African countries on four COVID-19 care centers (CCCs). The CCCs were set up in collaboration with a medical NGO with long experience in recording and monitoring data for cohorts and clinical trials in emergency contexts. The data were recorded using the WHO COVID-19 rapid core case report form.

ELIGIBILITY:
Inclusion Criteria:

* SARS-CoV-2 positive at RT-PCR

Exclusion Criteria:

* Asymptomatic patients

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: People hospitalized with symptomatic of COVID-19 and a positive RT-PCR SARS-CoV-2 test
Sampling Method: Non-Probability Sample
Enrollment: 2495 (Actual)
Dates: Start 2020-03-01 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-03-01 (Actual)

PRIMARY OUTCOMES:
Mortality | During hospitalization, with an average of 11 days
  In hospital mortality

SECONDARY OUTCOMES:
Clinical worsening | Hospitalization, with an average of 11 days
  Combination of an SpO2 <94% at least once during follow-up (including at baseline), use of oxygen therapy at any time during follow-up, or death

CONTACTS AND LOCATIONS:
Overall Officials: Denis Malvy, Pr, Principal Investigator — CHU Bordeaux, INSERM 1219
Locations (3):
- Burkina Faso (2):
  - Chu Tengandogo, Ouagadougou
  - Clinique Princesse Sarah, Ouagadougou
- Chu Donka, Conakry, Guinea

IPD SHARING:
Plan to Share IPD: Undecided